CLINICAL TRIAL: NCT04207983
Title: A 48 Week Phase II, Randomized, Open-Label, Multicenter, Study to Evaluate the Efficacy and Safety of Two (2) EYS606 Treatment Regimens in Subjects With Active Chronic Non-infectious Uveitis (CNIU)
Brief Title: A 48 Week Study to Evaluate the Efficacy and Safety of Two (2) EYS606 Treatment Regimens in Subjects With Active Chronic Non-infectious Uveitis (CNIU)
Acronym: ELECTRO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eyevensys (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EYS606-CT2
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Non-infectious Uveitis

STUDY DESIGN:
Intervention Model Description: Part I (Safety cohort phase) - no randomization will take place; subjects will be consecutively assigned to one of two sequential safety cohort Regimens and receive two administrations of EYS606
  Part II (Randomized comparison phase) - 1:1 randomization to either Treatment Arm A (Regimen 1 or 2 based upon recommendation by the DSMB, n=25) or Treatment Arm B (Regimen 3, n=25)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Treatment Arm A (Re-administration) (Experimental): Two administrations of EYS606 (135μg pEYS606/90 μL). The frequency between the two administrations will be determined by the DSMB upon completion of the Part I safety cohorts.
  Interventions: Combination Product: EYS606
- Treatment Arm B (Single administration) (Experimental): One administration of EYS606 (135μg pEYS606/90 μL) at the baseline visit (V1).
  Interventions: Combination Product: EYS606

INTERVENTIONS:
Combination Product: EYS606 — EYS606 is a DNA plasmid solution administered by electrotransfection into the ciliary muscle

SUMMARY:
The objective of the study is to evaluate the efficacy and safety of two different treatment regimens of EYS606.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, randomized open-label interventional study of EYS606 in subjects with active chronic non-infectious uveitis.

The maximum study duration per patient is 51 Weeks (including an up to 3 week screening period + 48 weeks follow-up after treatment).

The study will be conducted in 2 parts. Part I is a safety cohort phase that will enroll up to 6 subjects, Part II is the randomized comparison phase that will enroll up to an additional 50 subjects.

ELIGIBILITY:
Key Eligibility Criteria:

1. Subject must be 18 years of age or older.
2. Subject must have a diagnosis of chronic non-infectious uveitis of any anatomic subtype (anterior, intermediate, posterior or panuveitis).
3. Subject must have a history of chronic or recurrent non-infectious uveitis requiring or having required treatment with corticosteroids (systemic, periocular or intraocular) and/or systemic immunosuppressive medication(s) in the 12 months prior to the screening visit.
4. Best corrected visual acuity of

   * Study Part I: ≥ 5 and < 67 ETDRS letters in the study eye (equivalent to less than or equal to 20/50 but better than or equal to 20/800 Snellen).
   * Study Part II: ≥ 5 and < 77 ETDRS letters in the study eye (equivalent to less than or equal to 20/32 but better than or equal to 20/800 Snellen).
5. At the screening and baseline visits subject must have active chronic non-infectious uveitis as evidenced by at least one or more of the following in the study eye:

   * Active retinal vasculitis (retinal vascular leakage) involving the posterior pole confirmed by the reading center.
   * Vitreous haze grade ≥ 2+ (SUN classification).
   * Anterior chamber cell grade ≥ 2+ (SUN classification); anterior chamber cells must be present for subjects with a diagnosis of chronic anterior non-infectious uveitis.
   * Persistent macular edema (defined as central retinal thickness (CRT) > 300 microns or > 320 microns using Zeiss Cirrus and Topcon or Heidelberg Spectralis spectral domain ocular coherence tomography (SD-OCT) instruments, respectively) despite treatment with corticosteroids and/or immunosuppressive therapy for at least 4 weeks prior to screening.
6. Subject receiving concomitant topical and/or systemic corticosteroids or allowed systemic immunosuppressive medications must have maintained the same treatment regimen (dosage/frequency) for at least 2 weeks prior to the baseline (V1) visit, (if applicable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Time to rescue therapy between the two EYS606 treatment regimens | Week 24
  Assessment of efficacy measured as time to rescue therapy required after treatment with EYS606

SECONDARY OUTCOMES:
Proportion (%) of subjects responded to the treatment | Week 8 and 24
  Measured as an improvement in anterior cell grade and vitreous haze grade according to the SUN scale, retinal vessel leakage using fluorescein angiography, central retinal thickness using ocular coherence tomography, and an increase in visual acuity using EDTRS compared to baseline
Proportion (%) of subjects achieving and maintaining active chronic noninfectious posterior uveitis (CNIU) | Week 24
  Measured as an improvement in anterior cell grade and vitreous haze grade according to the SUN scale, retinal vessel leakage using fluorescein angiography, central retinal thickness using ocular coherence tomography, and an increase in visual acuity using EDTRS compared to baseline
Median time to control of active CNIU | Each Visit up to Week 48
  Measured as an improvement in anterior cell grade and vitreous haze grade according to the SUN scale, retinal vessel leakage using fluorescein angiography, and central retinal thickness using ocular coherence tomography
Median time to loss of treatment effect | Each Visit up to Week 48
  Measured as an worsening in anterior cell grade and vitreous haze grade according to the SUN scale, retinal vessel leakage using fluorescein angiography, central retinal thickness using ocular coherence tomography, decrease in visual acuity using EDTRS, and any increase in the frequency of dose of specified concomitant medications
Median change in visual acuity | Each Visit up to Week 48
  Measured in change from baseline in best-corrected visual acuity using EDTRS

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Texas Retina Associates, Arlington, Texas
  - Houston Eye Associates, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Touchard E, Benard R, Bigot K, Laffitte JD, Buggage R, Bordet T, Behar-Cohen F. Non-viral ocular gene therapy, pEYS606, for the treatment of non-infectious uveitis: Preclinical evaluation of the medicinal product. J Control Release. 2018 Sep 10;285:244-251. doi: 10.1016/j.jconrel.2018.07.013. Epub 2018 Aug 1. PMID 30009894